CLINICAL TRIAL: NCT00206635
Title: A Long-term Follow up of Patients Enrolled in the Pivotal Study of Betaseron® (Interferon Beta 1b) in Relapsing-remitting Multiple Sclerosis
Brief Title: Betaseron 16-Year Long-Term Follow-Up (LTF) in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare Pharmaceuticals Inc.
Other Study IDs: 308272
Record Dates: First submitted 2005-09-09; First posted 2005-09-21 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Betaseron was not administered as part of this study, only the treatment and disease status was assessed. As part of the MRI analysis Gadolinium was administered in patients who underwent this procedure

SUMMARY:
The purpose of this follow-up study is to look carefully at the long-term course of multiple sclerosis (MS) and possibly the long-term effects of Betaseron in the patients who were previously enrolled in the original North American study that led to the marketing approval of Betaseron.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients in North America have to have been previously enrolled in the original Betaseron trial from 1988-1993
* Be able to understand the consent form (or have a guardian who can)

Exclusion Criteria:

* North American patients cannot be included if they have not participated in the original Betaseron trial from 1988-1993

Min Age: 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Original pivotal trial population of Betaseron pivotal study (1989-1993)
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2005-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Description of long term course of disease | 16 years

SECONDARY OUTCOMES:
Comparison to natural history cohort | 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- United States (6):
  - Many Locations, Alabama
  - Many Locations, Arizona
  - Many Locations, California
  - Many Locations, Illinois
  - Many Locations, Maryland
  - Many Locations, Pennsylvania
- Canada (3):
  - Many Locations, British Columbia
  - Many Locations, Ontario
  - Many Locations, Quebec

REFERENCES:
- [Result] Ebers GC, Traboulsee A, Li D, Langdon D, Reder AT, Goodin DS, Bogumil T, Beckmann K, Wolf C, Konieczny A; Investigators of the 16-year Long-Term Follow-Up Study. Analysis of clinical outcomes according to original treatment groups 16 years after the pivotal IFNB-1b trial. J Neurol Neurosurg Psychiatry. 2010 Aug;81(8):907-12. doi: 10.1136/jnnp.2009.204123. Epub 2010 Jun 19. PMID 20562430
- [Result] Reder AT, Ebers GC, Traboulsee A, Li D, Langdon D, Goodin DS, Bogumil T, Beckmann K, Konieczny A; Investigators of the 16-Year Long-Term Follow-Up Study. Cross-sectional study assessing long-term safety of interferon-beta-1b for relapsing-remitting MS. Neurology. 2010 Jun 8;74(23):1877-85. doi: 10.1212/WNL.0b013e3181e240d0. PMID 20530324
- [Result] Goodin DS, Traboulsee A, Knappertz V, Reder AT, Li D, Langdon D, Wolf C, Beckmann K, Konieczny A, Ebers GC; 16-Year Long Term Follow-up Study Investigators. Relationship between early clinical characteristics and long term disability outcomes: 16 year cohort study (follow-up) of the pivotal interferon beta-1b trial in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2012 Mar;83(3):282-7. doi: 10.1136/jnnp-2011-301178. Epub 2011 Dec 21. PMID 22193561
- [Result] Goodin DS, Jones J, Li D, Traboulsee A, Reder AT, Beckmann K, Konieczny A, Knappertz V; 16-Year Long-Term Follow-up Study Investigators. Establishing long-term efficacy in chronic disease: use of recursive partitioning and propensity score adjustment to estimate outcome in MS. PLoS One. 2011;6(11):e22444. doi: 10.1371/journal.pone.0022444. Epub 2011 Nov 30. PMID 22140424